CLINICAL TRIAL: NCT02910089
Title: ENhancing Outcomes Through Goal Assessment and Generating Engagement in Diabetes Mellitus (ENGAGE-DM): A 12-month Study of the Impact of Combined Shared-decision Making and Brief Negotiated Interviewing on Disease Control and Medication Adherence in Patients With Diabetes
Brief Title: ENhancing Outcomes Through Goal Assessment and Generating Engagement in Diabetes Mellitus
Acronym: ENGAGE-DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Brigham Women's Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D1843R00254
Record Dates: First submitted 2016-08-04; First posted 2016-09-21 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shared Decision Making/Brief Negotiated Interviewing (Other): This prospective study will include 700 beneficiaries of Horizon Blue Cross Blue Shield of New Jersey (BCBSNJ).
  Interventions: Behavioral: Shared Decision Making
- Control Arm (No Intervention): Seven hundred patients will also be identified by Horizon Analytics as a control group for analyses purposes only; these patients will not be contacted.

INTERVENTIONS:
Behavioral: Shared Decision Making — This prospective study will include 700 beneficiaries of Horizon Blue Cross Blue Shield of New Jersey (BCBSNJ).
  Arms: Shared Decision Making/Brief Negotiated Interviewing

SUMMARY:
The purpose of this study is to evaluate whether a combination of pharmacist-delivered patient engagement techniques improves disease control and medication adherence among patients with poorly-controlled diabetes compared with usual care. These engagement techniques include shared decision-making and brief negotiated interviewing and are delivered telephonically.

DETAILED DESCRIPTION:
The US is facing a growing epidemic of type 2 diabetes. Among patients with poorly controlled diabetes, it is often not clear whether the problem is attributable to failure to appropriately intensify therapy, poor adherence to prescribed medications, unwillingness to accept new treatments or a combination of these factors. Multi-component pharmacist-delivered interventions, particularly those rooted in patient engagement, have been shown to be some of the most effective at improving adherence to chronic disease medications. Even though shared decision making and brief negotiated interviewing are complementary patient engagement techniques, the effectiveness of combining these 2 intervention approaches, especially in the management of diabetes, is unknown.

In this study of patients using at least one oral hypoglycemic therapy with poorly controlled disease, the investigators examine the impact of a shared decision making and behavioral interviewing intervention delivered telephonically by pharmacists, compared with usual care. Briefly, all patients allocated to the intervention will be mailed a patient decision aid to prime them for encounters with pharmacists. After receiving the decision aid, these patients will be asked to engage in and provide informed consent for at least 4 telephonic discussions with pharmacists about their diabetes treatment options, goals, and preferences, medication adherence, strategies for reducing adherence barriers, and the benefits of maintaining blood glucose control. The study is being conducted within a large insurer and consists of 700 patients each allocated to the intervention group and the control group. Analyses will be performed on an intent-to-treat basis.

After study completion, the investigators will also use predictive analytics to examine whether treatment response could be predicted based on patient characteristics, such as sociodemographic, clinical, medication use, and other motivational characteristics, which will provide information about which patients are most likely to benefit from the intervention.

ELIGIBILITY:
Inclusion:

* Commercially-insured beneficiaries
* Receive all medical/prescription drug benefits through Horizon
* On ≥1 one oral hypoglycemic agent
* Latest HbA1c measurement ≥ 8% (within previous 6 months)
* Provided phone number to Horizon

Exclusion:

- Currently using any insulin

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K. Choudhry, MD, Ph.D, Principal Investigator — Brigham Women's Health; Eric Wittbrodt, PharmD, MPH, Study Director — AstraZeneca
Locations (1):
- Research Site, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Lauffenburger JC, Ghazinouri R, Jan S, Makanji S, Ferro CA, Lewey J, Wittbrodt E, Lee J, Haff N, Fontanet CP, Choudhry NK. Impact of a novel pharmacist-delivered behavioral intervention for patients with poorly-controlled diabetes: The ENhancing outcomes through Goal Assessment and Generating Engagement in Diabetes Mellitus (ENGAGE-DM) pragmatic randomized trial. PLoS One. 2019 Apr 2;14(4):e0214754. doi: 10.1371/journal.pone.0214754. eCollection 2019. PMID 30939143
- See also: D1843R00254_ENGAGE_SAP_RedactedPDFA — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4399&filename=D1843R00254_ENGAGE_SAP_RedactedPDFA.pdf
- See also: D1843R00254_ENGAGE_Protocol_redactedPDFA — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4399&filename=D1843R00254_ENGAGE_DM_CSP_redacted_PDFA.pdf
- See also: D1843R00254_ENGAGE_SAP_RedactedPDFA — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4399&filename=D1843R00254_ENGAGE_SAP_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potentially eligible patients for inclusion in this study were those who: (1) were ≥18 years of age, (2) had filled a prescription for 1 or more oral hypoglycemic agents within the prior 12 months, and (3) had evidence of poor glycemic control (A1C ≥8%) within the previous 6 months.
Pre-assignment Details: Patients were excluded if, prior to identification, they had fewer than 3 months of continuous enrolment in the health plan, had recently filled insulin or had no available telephone contact information.
Period: Overall Study
Arm/Group | Shared Decision Making/Brief Negotiated Interviewing | Control Arm
Started (1,400 randomized patients) | 700 (Patients allocated to intervention) | 700 (Patients allocated to control)
Completed (38 patients (2.7%) were excluded from analysis because they lost insurance eligibility.) | 678 (22 patients ineligible (3.1%)) | 684 (16 Patients ineligible (2.3%))
Not Completed | 22 | 16
Not completed — Lost insurance eligibility | 22 | 16

BASELINE CHARACTERISTICS:
Population: Baseline Population excludes patients who lost insurance eligibility between the time of data pull and randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Shared Decision Making/Brief Negotiated Interviewing | Control Arm | Total
Number analyzed (Participants) | 678 | 684 | 1362
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Full Analysis Set
  Years | 55.0 (8.1) | 54.6 (8.4) | 54.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236 | 273 | 509
  Male | 442 | 411 | 853
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 678 | 684 | 1362

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Hemoglobin (HbA1c):
Description: Pre- to post-intervention change in mean HbA1c levels
Time Frame: baseline and at the end of 12 months post index date
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Shared Decision Making/Brief Negotiated Interviewing | Control Arm
Number analyzed (Participants) | 678 | 684
Percentage of HbA1c | -0.75 (1.96) | -0.79 (2.01)
Statistical Analysis 1: Comparison: Shared Decision Making/Brief Negotiated Interviewing vs Control Arm; Test type: Superiority — As per the SAP, no p-values were computed. Only point estimates with 95% confidence intervals were evaluated; GEE — As per the SAP, no p-values were computed. Only point estimates with 95% confidence intervals were evaluated; Generalized Estimating Equations with an identity link function (as a continuous variable) and normally distributed errors; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.2 to 0.32] — Model-based Mean Differences are reported that have been adjusted for imbalanced baseline characteristics

2. Secondary Outcome: Medication Adherence (PDC Measure)
Description: Mean Adherence (PDC) in each study arm in the follow-up period
Time Frame: during follow-up period of 12 months post index date
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Percentage of Days
Arm/Group | Shared Decision Making/Brief Negotiated Interviewing | Control Arm
Number analyzed (Participants) | 678 | 684
Percentage of Days | 67.5 (31.6) | 66.2 (32.7)
Statistical Analysis 1: Comparison: Shared Decision Making/Brief Negotiated Interviewing vs Control Arm; Average of the percentage (proportion x 100) of days covered across all subjects; Test type: Other; GEE — As per the SAP, no p-values were computed. Only point estimates with 95% confidence intervals were evaluated; Generalized Estimating Equations with an identity link function and normally distributed errors; Mean Difference (Final Values) = 1.00, 95% CI 2-sided [-2.42 to 4.40] — Model-based Mean Differences are reported that have been adjusted for imbalanced baseline characteristics

3. Secondary Outcome: Percentage (Proportion x 100) of Patients Achieving Optimal Adherence
Description: Percentage (Proportion x 100) of patients in each study arm achieving optimal adherence (PDC ≥0.80) in the follow-up period
Time Frame: during follow-up period of 12 months post index date
Population: Full Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Shared Decision Making/Brief Negotiated Interviewing | Control Arm
Number analyzed (Participants) | 678 | 684
Percentage of Participants | 46.2 | 45.0
Statistical Analysis 1: Comparison: Shared Decision Making/Brief Negotiated Interviewing vs Control Arm; Test type: Superiority; GEE — As per the SAP, no p-values were computed. Only point estimates with 95% confidence intervals were evaluated; Generalized Estimating Equations with a logit link and binary distributed errors; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.83 to 1.28]

4. Secondary Outcome: Patients Achieving HbA1c
Description: Percentage (Proportion x 100) of patients in each study arm achieving optimal HbA1c control in the follow-up period
Time Frame: baseline and at the end of 12 months post index date
Population: Full Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Shared Decision Making/Brief Negotiated Interviewing | Control Arm
Number analyzed (Participants) | 678 | 684
Percentage of Participants | 34.8 | 38.0
Statistical Analysis 1: Comparison: Shared Decision Making/Brief Negotiated Interviewing vs Control Arm; Test type: Other — As per the SAP, no p-values were computed. Only point estimates with 95% confidence intervals were evaluated; See comments — As per the SAP, no p-values were computed. Only point estimates with 95% confidence intervals were evaluated; Generalized Estimating Equations with a logit link and binary distributed errors; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.71 to 1.17]

ADVERSE EVENTS:
Time Frame: 12 months
Description: An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. In clinical studies, an AE can include an undesirable medical condition occurring at any time, including run-in or washout periods, even if no study treatment has been administered.
Arm/Group | Shared Decision Making/Brief Negotiated Interviewing | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/678 | 0/684
Serious Adverse Events (participants affected / at risk) | 5/678 | 0/684
Other Adverse Events (participants affected / at risk) | 1/678 | 0/684
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shared Decision Making/Brief Negotiated Interviewing (N=678) | Control Arm (N=684)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shared Decision Making/Brief Negotiated Interviewing (N=678) | Control Arm (N=684)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Evaluation of glycemic control is limited to participants who had baseline labs available. ~29% had missing outcomes data for the primary outcome; while we used multiple imputation to evaluate the study, this could have influenced the findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT02910089/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT02910089/SAP_001.pdf